CLINICAL TRIAL: NCT03860298
Title: A Phase I, Two-stage, and Open Label Study to Evaluate the Safety and Tolerability of Using NaviFUS System in Patients With Drug Resistant Epilepsy
Brief Title: Safety of Using NaviFUS System in Patients With Drug Resistant Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NaviFUS Corporation (Industry)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NF-2018-01
Record Dates: First submitted 2019-02-26; First posted 2019-03-01 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-06

CONDITIONS: Drug Resistant Epilepsy; Epilepsy, Drug Resistant; Drug Refractory Epilepsy; Epilepsy, Drug Refractory; Intractable Epilepsy; Epilepsy, Intractable; Medication Resistant Epilepsy; Refractory Epilepsy
Keywords: NaviFUS System; Focused Ultrasound; Drug Resistant Epilepsy; Intracranial Electroencephalography
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NaviFUS System (Experimental): FUS treatment for 10 minutes
  Interventions: Device: NaviFUS System

INTERVENTIONS:
Device: NaviFUS System — Using NaviFUS System treatment for 10 minutes in drug resistant epilepsy. The site of the NaviFUS exposure is where the future surgery will be removed. Patients will concomitant use of anti-epileptic drugs (AEDs).

SUMMARY:
This study is to evaluate the safety and the intracranial electroencephalography (iEEG) changes of using NaviFUS System for the treatment of patients with drug resistant epilepsy.

DETAILED DESCRIPTION:
This is a phase I, two-stage, prospective, open label, single center, and single-arm study. Eligible patients will be enrolled through the process of informed consent then will receive NaviFUS treatment one cycle. The time interval for each treatment cycle is 3 days, including baseline/treatment and 3 days observation. The site of the NaviFUS exposure is where the future surgery will be removed. Concomitantly use of anti-epileptic drugs (AEDs) will be monitored and recorded in the case report form (CRF). A total of six patients will be divided into two stages of recruitment, the first stage will recruit two patients, the second stage will be four patients. When the first stage is accomplished, the data and safety monitoring board (DSMB) will review the study data and provide the recommendations regarding continuation, termination, or other modifications of the study based on evaluation of observed adverse effects of the intervention. The second stage will begin to conduct after the DSMB agrees to proceed. In this clinical trial, stereo-electroencephalography (SEEG) exploration will be carried out during long-term video-EEG monitoring and excitability/irritability in focal epileptogenic region and epileptogenic network will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 20 years and older
2. Patients with drug resistant epilepsy (have failed treatment with at least two appropriate anti-epileptic drugs (AEDs) due to lack of efficacy) who hospitalized and underwent stereo-electroencephalography (SEEG) implantation for localization and delineation of epileptogenic focus for removing by surgery.
3. Seizure frequency is countable and available at least one month prior to study.
4. Willing and able to sign written informed consent and be able to comply with the study protocol for the duration of the study

Exclusion Criteria:

1. Patients with concurrent active psychiatric or mood disorders that in the opinion of the investigator would interfere with participation in the study
2. Patients have significant bleeding after SEEG implantation
3. Presence of pacemaker, implantable cardioverter-defibrillator (ICD), permanent medication pumps, cochlear implants, vagus nerve stimulation (VNS), or deep brain stimulation (DBS)
4. The skull bone area traversed by the sonication pathway is covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp
5. Clips or other metallic implanted objects in the FUS exposure path, except shunts
6. Abnormal coagulation profile: Platelet (PLT) < 100,000/μL, prothrombin time (PT) >14 sec or activated partial thromboplastin time (APTT) >36 sec, and international normalized ratio (INR) > 1.3
7. Pregnant or breast-feeding women
8. Coexisting medical problems of sufficient severity to limit compliance with the study
9. Known sensitivity/allergy to Magnetic Resonance Imaging (MRI) contrast agents or any of its components
10. Use of any recreational drugs or history of drug addiction or known history of substance or alcohol abuse
11. Patients has participated other clinical trial within 4 weeks of entering this study
12. Any other condition that, in the investigator's judgment, might affect study endpoints or might increase the risk to the patients or decrease the chance of obtaining satisfactory data needed to achieve the objectives of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability during study period using the NaviFUS System | 20 days
  The number and severity of adverse events

SECONDARY OUTCOMES:
Changes of iEEG | 3 days post FUS treatment
  Changes of excitability/irritability in focal epileptogenic region and epileptogenic network of iEEG at post FUS treatment by NaviFUS System from baseline period

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Yu Yu, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No